CLINICAL TRIAL: NCT01449916
Title: Improving Sepsis Diagnosis and Treatment: Simplified Severe Sepsis Protocol (SSSP)
Brief Title: Simplified Severe Sepsis Protocol in Zambia
Acronym: SSSP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: High mortality rate in intervention arm for patients with RR >40 AND SpO2 < 90%.
Sponsor: Vanderbilt University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSSP; R24TW007988 (NIH)
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Severe Sepsis
Keywords: Sepsis; Severe Sepsis; Protocol; Zambia
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simplified Severe Sepsis Protocol (Experimental): This protocol consists of an early aggressive fluid strategy, early blood cultures and antibiotics, and, when appropriate, blood transfusion and titratable dopamine. Monitoring is based on physical exam findings.
  Interventions: Other: Simplified Severe Sepsis Protocol
- Usual care (Active Comparator): Early blood cultures and antibiotics. Monitoring by study nurses as in experimental arm. Other interventions are according to admitting (non-study) doctors' orders.
  Interventions: Other: Simplified Severe Sepsis Protocol

INTERVENTIONS:
Other: Simplified Severe Sepsis Protocol — Early fluid protocol, early blood cultures and antibiotics; blood cultures and titrated dopamine in selected patients; monitoring based on vital signs and physical examination

SUMMARY:
This study is a randomized control trial assessing the impact of a simple evidence-based protocol for the treatment severe sepsis in Zambia. The intervention protocol consists of a scheduled fluid regimen, early blood culture and antibiotics, and dopamine and blood transfusion when necessary. It is hypothesized that the protocol will significantly decrease in-hospital mortality in patients with severe sepsis.

DETAILED DESCRIPTION:
In recent years, evidence-based protocols of bundled therapies have improved survival of severe sepsis in developed countries. However, in sub-Saharan Africa, simple therapies such as IV fluids and early antibiotics are frequently under-utilized. Furthermore, although tuberculosis is a common cause of severe sepsis in the region, accurate and timely diagnosis of tuberculosis-associated severe sepsis remains elusive.

The aims of this study are (1) To assess the impact on survival of a simple evidence-based protocol for severe sepsis, (2) To evaluate the cost of implementation for a simplified severe sepsis protocol (3) To develop a clinical diagnostic score for identifying tuberculosis in HIV positive patients with severe sepsis (4) To assess the performance of the Xpert TB/RIF rapid PCR system for diagnosing tuberculosis in HIV positive patients with severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Suspected infection
* 2 or more of SIRS criteria:

  * Heart rate >90/min
  * Respiratory rate >20/min
  * Temperature >= 38° C or <= 36° C
  * White blood count > 12,000 or < 4,000/µL
* 1 or more of the following signs of end-organ dysfunction

  * Systolic blood pressure < 90 mm Hg
  * Mean arterial blood pressure (MAP) < 65 mm Hg
  * Confusion/altered mentation
  * Urine output < 0.5 mL/kg/hr
  * Creatinine increase > 0.5 mg/dL
  * Creatinine > 0.5 mg/dL above upper limit of normal
  * Platelet < 100x109/L
  * Respiratory rate > 40/min
  * Jaundice

Exclusion Criteria:

* GI bleed
* Need for urgent surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
In-hospital all cause mortality | During hospitalization, expected average 14 days

SECONDARY OUTCOMES:
28-day all-cause mortality | 28-day
In-hospital all cause mortality adjusted for illness severity | During hospitalization, expected average 14 days
  Adjusted for SAPS3 score
28-day all cause mortality adjusted for baseline illness severity | 28-day
  Adjusted for SAPS3 score
Cumulative adverse events | During hospitalization, expected average 14 days
  A composite outcome consisting of dopamine extravasation, dopamine-associated tissue ischemia or necrosis, iatrogenic pulmonary oedema, and transfusion-related adverse events.
Treatment cost per patient | During hospitalization, expected average 14 days
  A budget impact analysis will determine the cost of treatment per patient using a mix of direct measurements and micro-cost observation.
Antibiotic changed due to culture results | During hospitalization, expected average 14 days
  The proportion of patients whose antibiotic regimen was changed due to information obtained from blood culture results.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Andrews, MD, Principal Investigator — Vanderbilt University and University of Zambia
Locations (1):
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No